CLINICAL TRIAL: NCT06351475
Title: Evaluation de l'efficacité du Remplissage Vasculaire Par de l'ALBUmine Humaine 20% + Ringer Lactate comparé au Ringer Lactate Seul Chez Les Patients opérés Par cytoréduction Avec CHimiothérapie Intrapéritonéale hyPerthermique
Brief Title: Efficacy of Intraoperative Use of 20% Albumin Combined With Ringer Lactate Versus Ringer Lactate During Cytoreductive Surgery With Hyperthermic Intraperitoneal Chemotherapy
Acronym: ALBUCHIP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: APHP230864
Record Dates: First submitted 2024-04-02; First posted 2024-04-08 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Peritoneal Neoplasms; Hyperthermic Intraperitoneal Chemotherapy; Intraoperative Care; Fluid Therapy; Postoperative Complications
Keywords: Cytoreductive surgery; Hyperthermic intraperitoneal chemotherapy; Albumin administration; Fluid therapy; Post operative prognosis; Randomized clinical trial; Open label clinical trial
MeSH Terms: conditions — Peritoneal Neoplasms; Postoperative Complications

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 20% Albumin + Ringer Lactate group (Experimental): Per-operative fluid therapy consisting in Ringer Lactate combined with 20% albumin. Patients will receive a bolus of 3 mL/kg on one hour of 20% albumin from anaesthetic induction. Then, infusion of 20% albumin (100 mL, 20g) will be administered for each 1200 mL of vascular filling by Ringer Lactate. Dosage of intra operative albuminemia will be realized 2 hours after the end of the bolus or infusion to ensure albuminemia is within the target concentrations (35-45 g/L). Use of 20% albumin will be realized for the entire duration of the surgery and stopped at the end of the surgery.
  Interventions: Other: Intra-operative albumin administration
- Control group (Active Comparator): Ringer Lactate for intra operative fluid management based on the latest scientific recommendations. As the the study is an open labelled randomized clinical trial, placebo use is not planned.
  Interventions: Other: Control

INTERVENTIONS:
Other: Intra-operative albumin administration — Patients randomized in the intervention group (20% albumin + Ringer Lactate) will receive, during cytoreductive surgery with HIPEC, fluid therapy consisting in Ringer Lactate (based on a fluid management protocol specifically set up for the study, and based on latest recommendations) combined with 20% albumin. Patients randomized in the intervention group will receive a bolus of 3 mL/kg on one hour of 20% albumin from anesthetic induction . Dosage of albuminemia will be done 2 hours after the end of the bolus (target of 35-45 g/L of intra operative albuminemia). Then, infusion of 20% albumin (100 mL, 20g) will be administered for each 1200 mL of vascular filling by Ringer Lactate. Dosage of intra operative albuminemia will be realized 2 hours after the end of the bolus or infusion to ensure albuminemia is within the target concentrations (35-45 g/L). Use of 20% albumin will be realized for the entire duration of the surgery and stopped at the end of the surgery.
  Arms: 20% Albumin + Ringer Lactate group
Other: Control — Ringer lactate
  Arms: Control group

SUMMARY:
Introduction Cytoreductive surgery (CRS) with hyperthermic intraperitoneal chemotherapy (HIPEC) is considered as the standard of care for the treatment of peritoneal metastases. Cytoreductive surgery with HIPEC is characterized by large intra operative fluid shift secondary to surgical resection, peritoneal inflammation and capillary shifts, requesting high volume of intra operative fluid therapy. Previous studies found a strong association between intra operative hypovolemia or volume overload with post operative outcomes. Albumin as an intravenous fluid has been widely studied in critical ill patients, but evaluation of its efficacy during major surgery on post operative clinical outcomes are lacking. We hypothesize that a reduction of intra operative crystalloid volume infusion by using 20% albumin during CRS with HIPEC could improve patients' prognosis. The aim of this study will be to assess the efficacy of 20% albumin combined with Ringer Lactate versus Ringer Lactate for fluid therapy during CRS with HIPEC on post operative outcome at 28 day.

Methods and analysis The study protocol has been designed and written in accordance with the Prospective randomised, comparative, controlled, prospective, open-label, with parallel group and multicentre clinical trial.

Recruitment, randomisation and allocation Information on the study and screening of patients will be conducted during the consultation of anaesthesia (= selection visit), 2 months at 3 days before the surgery. Information notice and consent form will be delivered. The day before the surgery, anaesthesiologist who will conduct the pre anaesthetic visit will be able to include patients in the study (=inclusion visit). Randomisation will be done at the inclusion visit after information and signature of consent form of voluntary patients. A randomization number will be assigned. The 1:1 randomisation will be centralized via an online interface ensuring secret group assignment, and based on predefined randomisation lists with variable-size permutation blocks, stratified by center. Randomisation will be accomplished using a computer-generated random sequence.

Randomized Open, Blinded endpoint (PROBE) design. This study is a randomised, comparative, controlled, prospective, open-label, with parallel group and multicentre clinical trial.

Intervention

* 20% Albumin + Ringer Lactate group (intervention group) Per-operative fluid therapy consisting in Ringer Lactate combined with 20% albumin. Patients will receive a bolus of 3 mL/kg on one hour of 20% albumin from anaesthetic induction. Then, infusion of 20% albumin (100 mL, 20g) will be administered for each 1200 mL of vascular filling by Ringer Lactate. Dosage of intra operative albuminemia will be realized 2 hours after the end of the bolus or infusion to ensure albuminemia is within the target concentrations (35-45 g/L). Use of 20% albumin will be realized for the entire duration of the surgery and stopped at the end of the surgery.
* Control group Ringer Lactate for intra operative fluid management based on the latest scientific recommendations. As the the study is an open labelled randomized clinical trial, placebo use is not planned.

Outcome measures The primary outcome will be the Comprehensive Complication Index (CCI score) at day 28 after CRS with HIPEC. Secondary outcomes are mortality at day 28, CCI score at day 7, volume of intra operative and post operative (48h) post operative fluid therapy, cumulated incidence of surgical post operative complications, cumulated incidence of medical post operative complications, need for mechanical ventilation, renal replacement therapy between surgery and day 28, SOFA score variation between pre operative period and 48h after surgery, number of days alive out of intensive care unit and out of hospital until day 28

Sample size calculation To ensure a power of 80%, a number of patients 130 (65 patients by group) will be necessary with a reduction of 13.6 (SD 24) points of the CCI score at day 28 in the intervention group. Because of a risk of neoplastic evolution between anaesthetic consultation and randomisation (10% of early cancellation), a total of 146 patients (73 by group) will be included in the study.

Discussion In summary, ALBUCHIP study will be the first randomized clinical trial assessing efficacy of intraoperative use of 20% albumin combined with Ringer Lactate versus Ringer Lactate during CRS with HIPEC. Results yielded from this study will be helpful for vascular filling during CRS with HIPEC but, thanks to ancillary studies, to improve pathophysiological understanding of this surgery.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 18 years old and older
* Planned cytoreductive surgery with HIPEC for peritoneal carcinomatosis (from gynaecological or digestive origin)
* Patient volunteer for the study and provided written informed consent
* Patient affiliated to the French Health Insurance

Exclusion Criteria:

* Adults >75 years old
* Functional status rendering the patient ineligible for cytoreduction with CHIP (ECOG > 2 or Karnofsky index < 75)
* Pre-existing preoperative conditions affecting albuminemia (hepatic cirrhosis, nephrotic syndrome, exudative enteropathy, malnutrition)
* Severe preoperative hypoalbuminemia (albuminemia < 20 g/L)
* History of chronic left heart failure with reduced left ventricular ejection fraction (left ventricular ejection fraction < 40%)
* Patients at high risk of perioperative and postoperative pulmonary complications (atelectasis, significant pleural effusions)
* Significant ascites with preoperative respiratory repercussions
* Uncontrolled diabetes (HbA1c > 8.5%)
* Allergy to exogenous human albumin and its excipients.
* Contraindication to the administration of Ringer's lactate (history of allergy)
* Hyperkalemia > 6.0 mmol/L
* Hypercalcemia (total calcium > 2.60 mmol/L)
* Chronic use of digitalis and hyperkalemic diuretics
* Pregnancy, breastfeeding
* Known preoperative renal failure (GFR < 30 mL/min/1.73m2 or extrarenal purification)
* Recent brain trauma < 6 months (traumatic, ischemic, or hemorrhagic)
* Participation in another interventional study involving human subjects or being in the exclusion period following a previous study involving human subjects, if applicable
* Patient deprived of liberty
* Patient under guardianship or curatorship

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-09-03 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Comprehensive Complication Index score | At day 28
  The Comprehensive Complication Index (CCI) is a score ranging from 0 to 100, calculated using all complications and their treatment after abdominal surgery.
  The CCI is that it is a linear scale ranging from 0 to 100, where 100 represents death

SECONDARY OUTCOMES:
Comprehensive Complication Index score | At day 7
  The Comprehensive Complication Index (CCI) is a score ranging from 0 to 100, calculated using all complications and their treatment after abdominal surgery.
  The CCI is that it is a linear scale ranging from 0 to 100, where 100 represents death
Volume of intra operative and post operative fluid therapy | 48 hours after surgery
Cumulative incidence of surgical post operative complications | Up to day 28
Incidence of infectious complications | Up to day 28
Number of days under mechanical ventilation outside the operating room | Up to day 28
  Between surgery and day 28
Number of days under renal replacement therapy | Up to day 28
  Between surgery and day 28
Sequential organ failure assessment (SOFA) score variation | 48 hours after surgery
  Between pre operative period and 48h after surgery
Number of days alive out of intensive care unit | Up to day 28
Number of days alive out of hospital | Up to day 28
Incidence of medical complications | Up to day 28
Cumulative incidence of death in intensive care unit | Up to day 28
Cumulative incidence of death in hospital | Up to day 28
SOFA score | At day 28
  Sequential Organ Failure Assessment Score varies from 0 to 4 and permit to assess organ failure. A higher score indicates better neurological function
Number of days under vasopressors | Up to day 28
Proportion of patients with allergic complications to albumin | At day 133

CONTACTS AND LOCATIONS:
Locations (7):
- France (7):
  - Institut régional du Cancer de Montpellier, Montpellier
  - La Pitié Salpetriere hospital, Paris
  - Lariboisière hospital, Paris
  - Saint Louis hospital, Paris
  - Robert Debré hospital, Reims
  - Hôpital Hautepierre / UIC ARMO, Strasbourg
  - Gustave Roussy Institute, Villejuif

IPD SHARING:
Plan to Share IPD: Undecided